CLINICAL TRIAL: NCT02588729
Title: A Mobile Smartphone Application to Promote a Healthy Diet and Physical Activity Among Pregnant Women With Gestational Diabetes Mellitus - RCT
Brief Title: A Mobile Smartphone Application to Promote a Healthy Diet and Physical Activity Among Pregnant Women With GDM - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Universitetssenteret på Kjeller (Other); Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other); University Hospital, Akershus (Other); The Norwegian Centre for Minority Health Research (Other)
Responsible Party: Principal Investigator, Mirjam Lukasse, Associate professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 38942
Record Dates: First submitted 2015-08-31; First posted 2015-10-28 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes; app; RCT; diet; physical activity
MeSH Terms: conditions — Diabetes, Gestational; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregnant+ app for smartphone (Gravid+) (Experimental): The intervention consists of the Pregnant+app downloaded on women's smartphone. The app contains culturally adapted information about physical activity, diet and management of GDM. The Gravid+app will be available in Norwegain, Urdu and Somali. Women will have the opportunity to automatically transfer their blood glucose levels to their smartphones via Bluetooth.
  Interventions: Other: Pregnant+ app for smartphone
- No admission to Pregnant+ app (Gravid+) (No Intervention): The control group will receive standard care at the outpatient departments. Participants to not receive the Pregnancy

INTERVENTIONS:
Other: Pregnant+ app for smartphone — The Pregnant+app for smartphone with information about a healthy diet, physical activity and management of gestational diabetes mellitus.
  Arms: Pregnant+ app for smartphone (Gravid+)

SUMMARY:
In this study, the investigators will test a new way to communicate advice on diet and lifestyle to women with gestational diabetes mellitus by app downloaded on women's smartphone. The app wishes to motivate women to have a healthy diet, and be physically active. It allows automatic transfer of blood glucose measures from the glucose meter to the smartphone. The women will answer questionnaires during pregnancy and be followed up three months postpartum.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM), diabetes occuring for the first time during pregnancy, is an increasing problem worldwide. It may affect both the woman's and their offspring's health. Women with GDM have an increased risk of developing type 2 diabetes later in life. Pregnancy, offers a window of opportunity to instigate lasting changes beneficial for them and their families. Considering new technology available and used by women generally, new methods to communicate lifestyle and dietary advice are required.

The present study, a multi-center, randomised controlled trial includes five outpatients clinics in the greater Oslo Region and will include 230 pregnant women with gestational diabets mellitus. Data will be collected by three questionnaires during the study period, one at entry, before 33+0 weeks of gestation, one at 36 weeks and the last questionnaire at around three months postpartum. During pregnancy, the questionniares will be answered using an iPad while the last questionnaire will be on a website or through an interview.

Additional information will be collected from the women's medical record.

The intervention in this study is an app, called the Pregnant+ app (Gravid+) for smartphone. The app aims to reach women who are fluent in either Norwegian, Urdu or Somali. It has been translated from Norwegian and culturally adapted to women speaking Urdu or Somali. Women participating in the study can choose between different food cultures and they can set their personal lifestyle goals. Information about gestational diabetes, psysical activity, diet and food recipes are provided in the app. Half of the women in this study, will be given the app, downloaded on their smartphone.The opportunity to automatically transfer bloodglucose measures to the smartphone, presented in either a list or a graph, gives women an overview and therefore easier controll over their glucose levels.

The intervention will take place in the ordinary consultation at the outpatient clinics and no extra consultation are needed.

The data will be analysed according to intention to treat methods and with a parcicipatin rate on 75% it will take approximately 20 months to recruite 230 pregnant women. To detect a differences of 10% between the intervention group and the control group, 115 women are required in each group.

The Regional Committees for Medical and Health Research Ethics South East, (REK) reviewed the investigators' application and deemed ethical approval not required as the investigators' study does not test new medication or treatment, nor seeks to find new information about GDM but only tests a new way of communicating known and approved lifestyle advice to women with GDM.

For each hospital the investigators received approval from the appropriate Board for patient privacy protection (PVO: Personvernombud). The study was approved at each hospital by the responsible medical officer.

The investigators' study has been approved by the Norwegian Social Science Data Services.

The RCT will be published in an international peer-reviewed scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* First visit with gestational diabetes in this pregnancy
* Has her own smartphone
* Pregnancy up to 32 weeks and 6 days of gestation
* Fluent in Norwegian, Urdu or Somali
* Aged 18 years old and older

Exclusion Criteria:

* Pregnant with more than one fetus
* Lactose or gluten intolerance
* Known type 1 diabetes (insulin dependent)
* Known type 2 diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test (OGTT), fasting and 2 hours blood glucose level after intake up til 75gr glucose (1.75gr/kg body weight) | Approximately three months after delivery.
  Part of routine care for women who had GDM, is an OGTT about three months postpartum, taken at their laboratory and reported to the investigators.Number of participants with level below 7.5 mmol

SECONDARY OUTCOMES:
complications of pregnancy | Data will be collected prior to 33 weeks gestation, at 36 weeks gestation and up to 4 months postpartum
  Raised BP, vaginal bleeding, amniotic fluid leakage, preeclampsia, nausea and vomitting, Braxton Hicks Contractions, UTI, Candida vaginal infection, pelvic girdle pain
Dietary intake measured by "Fit for fødsel Food questionnaire" | Data will be collected prior to 33 weeks gestation, at 36 weeks gestation and up to 4 months postpartum
  Fit for fødsel Food questionnaire, 41 questions. Number of participants following ten items of advice on low glucose, high fiber diet.
Knowledge of gestational diabetes | Data will be collected prior to 33 weeks gestation, and at 36 weeks gestation
  7 questions assessing knowledge of gestational diabetes and understanding of glucose measurements and control of those. Number of participants with high understanding of GDM at 36 weeks, and number of participants with increasing knowledge.
Physical activity | Data wil be collected prior to 33 weeks gestation, at 36 weeks gestation, up to 4 months postpartum
  PPAQ:Pregnancy Physical Activity Questionnaire (37 questions). Comparison of participants in both arms of the study for Level of physical activity.
  Number of participants with low, moderate or high level of activity.
Depression | Data will be collected prior to 33 weeks gestation, at 36 weeks gestation, up to 4 months postpartum
  Edinburgh Depression Scale- short version, 5 questions. Number of participants with depression. Cut-off at either total score of 7 or 8.
Motivation for physical activity | Data will be collected prior to 33 weeks gestation, at 36 weeks gestation, up to 4 months postpartum
  4 questions assessing women's motivation to be physically active, number of women with high score and increasing score.
Motivation for eating healthy | Data will be collected prior to 33 weeks gestation, at 36 weeks, up to 4 months postpartum
  3 questions assessing women's motivation to eat healthy, number of women with high score and increasing score.
Mode of delivery and complications at birth for the mother | at birth
  From the Medical records, number of women for each group: induction, mode of delivery, shoulderdystocia, postpartum haemorrhage, Sphincter rupture, episiotomi, manual removal of placenta, Hb below 11 gr/dl, infection, removal of retained products.
Complications for the newborn | at birth
  Number of newborns who were transferred to intensive care unit, who were diagnosed with hypoglycaemia, information from the Medical records.
Condition of the newborn | at birth and approx three months postpartum
  Number of newborns with Apgar score below 7 at 5 minutes, birth weight above different cut-offs (3.5 kg and 4kg), full breastfeeding and other nutrition from pasient notes and 3 months postpartum questionnaire.
Starting medication for controlling blood glucose levels for the pregnant woman | during pregnancy
  Number of patients who start to use insulin or Metformin during pregnancy, information from the patient notes
Blood glucose control during pregnancy | during pregnancy
  Number of patients with, fasting glucose over 5.5 gr/dl, HbA1c above 7.0% at 30,32,34,36,38 and 40 weeks
HbA1c | Approx three months postpartum
  Measured at home by visiting researcher, finger prick blood.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Lukasse, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo university hospital, Oslo, Norway

REFERENCES:
- [Background] Garnweidner-Holme LM, Borgen I, Garitano I, Noll J, Lukasse M. Designing and Developing a Mobile Smartphone Application for Women with Gestational Diabetes Mellitus Followed-Up at Diabetes Outpatient Clinics in Norway. Healthcare (Basel). 2015 May 21;3(2):310-23. doi: 10.3390/healthcare3020310. PMID 27417764
- [Derived] Garnweidner-Holme L, Henriksen L, Bjerkan K, Lium J, Lukasse M. Factors associated with the level of physical activity in a multi-ethnic pregnant population - a cross-sectional study at the time of diagnosis with gestational diabetes. BMC Pregnancy Childbirth. 2022 Jan 3;22(1):1. doi: 10.1186/s12884-021-04335-x. PMID 34979996
- [Derived] Garnweidner-Holme L, Henriksen L, Torheim LE, Lukasse M. Effect of the Pregnant+ Smartphone App on the Dietary Behavior of Women With Gestational Diabetes Mellitus: Secondary Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 4;8(11):e18614. doi: 10.2196/18614. PMID 33146620
- [Derived] Borgen I, Smastuen MC, Jacobsen AF, Garnweidner-Holme LM, Fayyad S, Noll J, Lukasse M. Effect of the Pregnant+ smartphone application in women with gestational diabetes mellitus: a randomised controlled trial in Norway. BMJ Open. 2019 Nov 11;9(11):e030884. doi: 10.1136/bmjopen-2019-030884. PMID 31719080
- [Derived] Borgen I, Garnweidner-Holme LM, Jacobsen AF, Bjerkan K, Fayyad S, Joranger P, Lilleengen AM, Mosdol A, Noll J, Smastuen MC, Terragni L, Torheim LE, Lukasse M. Smartphone application for women with gestational diabetes mellitus: a study protocol for a multicentre randomised controlled trial. BMJ Open. 2017 Mar 27;7(3):e013117. doi: 10.1136/bmjopen-2016-013117. PMID 28348183